CLINICAL TRIAL: NCT04006444
Title: Characterization of the Iatrogenic Drug Risk in Elderly Patients With Chronic Pain Who Consult the Pain Assessment and Treatment Centre at the Nimes University Hospital
Acronym: ALGOGER
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: Local/2017/GL-01
Record Dates: First submitted 2019-07-01; First posted 2019-07-05 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2019-06

CONDITIONS: Iatrogenic Drug Risk; Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Chronic pain may be an additional risk factor for drug iatrogeny due to its management and also drug non-compliance in the geriatric population.

it seems interesting to carry out an inventory of the iatrogenic risk before and after the consultation at the pain centre to enable us to identify the patients most at risk. This study would make it possible to characterize elderly patients with chronic pain, in order to consider, in a future study, setting up a pharmaceutical consultation.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be affiliated or beneficiary of a health insurance
* Patient ≥ 65 years old
* Having an outpatient consultation at the pain centre of the Nîmes University hospital of for chronic pain
* Available for pharmaceutical consultation about 30 minutes

Exclusion Criteria:

* It is impossible to give information
* The patient objects to participating in this study

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: patients aged at least 65 years consulting at the pain centre of the Nîmes University Hospital for chronic pain
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-06-16 (Actual); Study Completion 2018-06-16 (Actual)

PRIMARY OUTCOMES:
Evolution of the ADE Geriatric risk score | 2018
  The score is calculated on 10 points based on 3 criteria : number of drugs prescribed, prescription of neuroleptics and the initiation of an anticoagulant prescription less than 3 months old. It classifies patients into 3 risk categories: a low risk level for a score of 0 to 1 point, a medium risk level for a score of 2 to 5 points and a high risk level for a score of 6 to 10 points.

SECONDARY OUTCOMES:
rate of patients with a low, medium or high risk level calculated by ADE Geriatric risk score according to the type of pain | 2018
  The score is calculated on 10 points based on 3 criteria : number of drugs prescribed, prescription of neuroleptics and the initiation of an anticoagulant prescription less than 3 months old. It classifies patients into 3 risk categories: a low risk level for a score of 0 to 1 point, a medium risk level for a score of 2 to 5 points and a high risk level for a score of 6 to 10 points.

CONTACTS AND LOCATIONS:
Overall Officials: geraldine leguelinel, Dr, Principal Investigator — CHU NIMES
Locations (1):
- CHU Nimes, Nîmes, France

REFERENCES:
- [Derived] Jambon J, Choukroun C, Roux-Marson C, Viel E, Leguelinel-Blache G. What Is the Medication Iatrogenic Risk in Elderly Outpatients for Chronic Pain? Clin Neuropharmacol. 2022 May-Jun 01;45(3):65-71. doi: 10.1097/WNF.0000000000000505. PMID 35579486